CLINICAL TRIAL: NCT05728775
Title: REmimazolam vs Propofol Total Intravenous Anesthesia on Outcomes After Major Noncardiac SurgEry (REPOSE-2): A Multicenter Randomized Controlled Trial
Brief Title: REmimazolam vs Propofol Total Intravenous Anesthesia on Outcomes After Major Noncardiac SurgEry
Acronym: REPOSE-2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NFEC-2022-286
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Anesthesia; Surgery-Complications
MeSH Terms: interventions — remimazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam TIVA (Experimental): Remimazolam is administered at 6-12 mg/kg/h intravenously for anesthesia induction and at 1.0-2.0 mg/kg/h for maintenance of general anesthesia. The dose is titrated to maintain Bispectral Index value between 40 and 60.
  Interventions: Drug: Remimazolam
- Propofol TIVA (Active Comparator): Propofol 1.5-2.5mg/kg is administered intravenously for anesthesia induction and propofol at 4-12mg/kg/h is used for maintenance of general anesthesia. The dose is titrated to maintain Bispectral Index value between 40 and 60.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is administered intravenously for induction and maintenance of general anesthesia.
  Arms: Remimazolam TIVA
Drug: Propofol — Propofol is administered intravenously for induction and maintenance of general anesthesia.
  Arms: Propofol TIVA

SUMMARY:
The goal of this randomized controlled trial is to compare total intravenous anesthesia with remimazolam vs total intravenous anesthesia with propofol in moderate-to-high risk patients undergoing major elective noncardiac surgery under general anesthesia. The primary hypothesis is that total intravenous anesthesia with remimazolam can increase days alive and out of hospital at postoperative day 30 compared with total intravenous anesthesia with propofol.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥45 years;
* Undergoing elective major surgery under general anesthesia (expected surgery time >2 h, expected length of postoperative stay >2 d);
* Fulfilling ≥1 of the following criteria:

  1. history of coronary artery disease;
  2. history of stroke;
  3. history of congestive heart failure;
  4. preoperative NT-proBNP >200 pg/mL or BNP>92 pg/mL;
  5. age ≥70 years;
  6. diabetes requiring medical treatment;
  7. ASA status 3 or 4;
  8. history of chronic kidney disease (preoperative sCr >133 μmol/L or 1.5 mg/dL);
  9. history of peripheral arterial disease;
  10. preoperative serum albumin <30 g/L;
  11. preoperative hemoglobin <100 g/L.

Exclusion Criteria:

* Undergoing organ transplantation, cardiac, craniocerebral, burn or interventional operations;
* Low risk or minor surgery
* End-stage renal disease requiring renal-replacement therapy;
* Hepatic dysfunction (Child B or C);
* Previous liver or kidney transplantation;
* Previous allergy to general anesthetics;
* Unable to receive bispectral index monitoring;
* ASA score ≥5;
* Exposure to general anesthesia in prior 30 days or anticipated re-exposure to general anesthesia within 30 days after surgery;
* Need for prolonged airway protection or mechanical ventilatory support after surgery;
* Current participation in another interventional study;
* Previous participation in this study;
* Pregnant or breastfeeding women.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7188 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Days alive and out of hospital at day 30 | 30 days after randomization
  Number of days alive and out of hospital

SECONDARY OUTCOMES:
All-cause 30-day mortality | 30 days after randomization
  Number of patients who die of any cause
Length of hospital stay | 30 days after randomization
  Number of days in hospital
Unplanned re-hospitalization | 30 days after randomization
  Number of patients who experience unplanned hospital re-admissions
Postoperative complications | 30 days after randomization
  Number of patients who experience postoperative complications
Quality of Recovery-15 score on the first day after surgery | Postoperative day 1
  Using Quality of Recovery-15 questionnaire to evaluate the quality of perioperative recovery. Quality of Recovery-15 consists of 15 comprehensive questions, including physical comfort (5 items), psychological support (2 items), physical independence (2 items), emotional state (4 items), and pain (2 items), each item is scored with 0-10 points, 0 represents poor state, 10 represents good state, and the total score is the Quality of Recovery-15 score of the patient.

OTHER OUTCOMES:
Cancer recurrence | 3 years after randomization
  Number of patients who experience cancer recurrence after radical resection of cancer
All-cause 3-year mortality | 3 years after randomization
  Number of patients who die of any cause

CONTACTS AND LOCATIONS:
Locations (44):
- China (44):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Huainanchaoyang Hospital, Huainan, Anhui
  - Suzhou First People's Hospital, Suzhou, Anhui
  - Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Xinqiao Hospital of Chongqing, Chongqing, Chongqing Municipality
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Southern Medical University Zhujiang Hospital, Guangzhou, Guangdong
  - Southern Medical University Nanfang Hospital, Guangzhou, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Qiandongnanzhou People's Hospital, Kaili, Guizhou
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Kaifeng Central Hospital, Kaifeng, Henan
  - The 989 Hospital of the People's Liberation Army Joint Support Force, Pingdingshan, Henan
  - Shangqiu Third People's Hospital, Shangqiu, Henan
  - Changge people's hospital, Xuchang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Henan Province Hospital of TCM, Zhengzhou, Henan
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan University People's Hospital, Wuhan, Hubei
  - The Central Hospital of Wuhan, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Hunan Provincial People's Hospital (The First Affiliated Hospital of Hunan Normal University), Changsha, Hunan
  - The First Affiliated Hospital Of University Of South China, Hengyang, Hunan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - The Second Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - The Second Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - General Hospital of Northern Theater Command, Shenyang, Liaoning
  - The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital, Jinan, Shandong
  - The 960th Hospital of the PLA Joint Logistic Support Force, Zibo, Shandong
  - Bao Ji City People's Hospital（BaoJi Emergency Medical Center）, Baoji, Shanxi
  - Fenyang Hospital of Shanxi Province, Fenyang, Shanxi
  - The First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Taiyuan, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Chongqing Western Hospital, Chongqing
  - Liangjiang Hospital of Chongqing Medical University, Chongqing

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: One year after the main trial result is published.